CLINICAL TRIAL: NCT01505452
Title: Translational Error in Flexion-extension Gap Balancing With Singe Radius Total Knee Arthroplasty
Brief Title: Study of Surgical Technique With Use of Single-radius Prosthesis in Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Athens Orthopedic Clinic, P.A. (Other)
Collaborators: Stryker Orthopaedics (Industry)
Responsible Party: Principal Investigator, Ormonde M. Mahoney, MD, Principal Investigator, Athens Orthopedic Clinic, P.A.
Other Study IDs: AOC-OM-Stryker-2009-0019
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Arthritis of Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to clinically demonstrate a phenomenon of measurement error that can occur during placement of a specific type of total knee replacement prosthesis (single radius femoral component) using a certain type of surgical technique (flexion/extension gap balancing).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo primary total knee arthroplasty performed by the principal investigator
* Use of a single radius posterior-stabilized TKA prosthesis is planned
* Spinal anesthetic is planned
* Diagnosis of osteoarthritis
* Has normal knee ligaments with no history of previous injury or surgery to ligaments, or other pathologic condition
* Has at least 100 degrees knee flexion preoperatively (measured by long goniometer)
* Gives valid informed consent
* Age 18 years or older

Exclusion Criteria:

* Patient receives general anesthetic
* Diagnosis other than osteoarthritis (e.g., rheumatoid arthritis, avascular necrosis, post-traumatic arthritis)
* History of any prior knee ligament injury, or any surgery to ligaments
* Any connective tissue disease affecting integrity of the ligaments (must have normal ligaments)
* History of long bone fracture in the affected leg
* Flexion contracture that would interfere with ability to establish extension gap reliably (judgment of investigator)
* Maximum pre-operative knee flexion is less than 100 degrees.
* Patient is non-ambulatory
* Any preclusion or inability to use navigation
* Treatment with single radius posterior stabilized TKA prosthesis is not indicated
* Participation is not in best interest of patient for any reason
* Cannot or does not give valid informed consent
* Female patient who is currently pregnant
* Age less than 18 years
* Body mass index greater than 40 kg/(m*m)
* Incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic based population (patients undergoing total knee replacement at an orthopedic surgery clinic).
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Difference in varus/vagus laxity of the knee joint measured with the knee positioned at a 90 degree angle with posteriorly stabilized vs. cruciate retaining trails in place. | At the time of the surgical procedure
  During the surgical procedure each participant will undergo measurement of varus/valgus laxity (in degrees) at 90 degrees knee flexion using both types of trial implants in sequence. We will evaluate whether the difference of varus/valgus laxity between the two surgical conditions is correlated to change in anterior/posterior relative position of the tibia (relative to femur) measured between the two conditions. A positive correlation between these two variables (change of position to change of laxity) would demonstrate a potential for measurement error that could occur during surgical procedures if position change of the tibia is not accounted for. All outcomes for this study are measured during the surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ormonde M Mahoney, MD, Principal Investigator — Athens Orthopedic Clinic
Locations (2):
- United States (2):
  - Athens Orthopedic Clinic, Athens, Georgia
  - St Mary's Hospital, Athens, Georgia